CLINICAL TRIAL: NCT02500862
Title: Characterization of Potential Biomarkers of Eye Disease and Vision Loss.
Brief Title: Characterization of Potential Biomarkers of Eye Disease and Vision
Acronym: EYE-MARKER
Status: Active, not recruiting | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: 4C-2015-08
Record Dates: First submitted 2015-07-10; First posted 2015-07-17 (Estimated); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Eye Disease
Keywords: Eye; Imaging
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Characterize potential biomarkers of sight-threatening eye diseases based on the information acquired in clinical practice at CEC, AIBILI

DETAILED DESCRIPTION:
This is a registry study. Only patients followed under the clinical practice at AIBILI Clinical Trial Centre, and with a signed informed consent form will be included.

Based on the clinical information collected under the clinical practice, and based on patients' characteristics, scientific questions will be raised and data will be collected and analysed accordingly.

Any procedure performed under clinical practice that may allow for the characterization of the disease and/or for the identification of potential biomarkers will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Any patient followed under the normal clinical practice at AIBILI Clinical Trial Centre, and with a AIBILI signed informed consent form for data collection, Imp. 11-7-2 "Consentimento Informado para tratamento de dados".

Exclusion criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any patient followed under the normal clinical practice at AIBILI Clinical Trial Centre, and with a AIBILI signed informed consent form for data collection, Imp. 11-7-2 "Consentimento Informado para tratamento de dados".
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Characterize potential biomarkers of sight-threatening eye diseases based on the information acquired in clinical practice at CEC, AIBILI. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Ribeiro, MsC, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- CEC, Coimbra, Portugal